

# Statistical Analysis Plan Cover Page

**Document Title:** Statistical Analysis Plan for Protocol PRO 140 CD 02-Extension

Protocol Number: PRO 140 CD 02-Extension

Protocol Title: An Extension Protocol for Subjects who Successfully Completed PRO140\_CD02

or PRO140 CD02 Open Label Study

Version: 4.0

**Document Date: 19-May-2020** 

NCT Number: NCT02990858



# STATISTICAL ANALYSIS PLAN FOR PROTOCOL PRO 140\_CD 02-EXTENSION

Sponsor:

CytoDyn

CytoDyn, Inc.

1111 Main Street, Suite 660 Vancouver, Washington

98660

(360) 980-8524-Work

(360) 980-8549-Fax

www.cytodyn.com

Protocol Number:

PRO 140 CD 02-Extension

**Protocol Title:** 

An Extension Protocol for Subjects who Successfully

Completed PRO140 CD02 or PRO140 CD02 Open Label

Study

**Protocol Date / Version:** 4.0/13-May-2019

**SAP Author:** 

Telephone:

Facsimile:

**Plan Version:** Version 0.2

Plan Date: 19May2020

| <b>Protocol Number:</b> | PRO 140_CD 02-Extension | |
|---|---|---|
| Protocol<br>Version/Date: | 4.0/ 13-May-2019 | |
| Protocol Name: | Protocol Name: An Extension Protocol for Subjects who Successfully Completed PRO140_CD02 or PRO140_CD02_Open Label Study | |
| Sponsor: | CytoDyn, Inc. 1111 Main Street, Suite 660 Vancouver, Washington 98660 | |
| Prepared by: | | |
| SAP Version: | Version 0.2 | 1 0.2 |
| SAP Date: | 19May2020 | |
| I have read and approve content: | the Statistical Analysis Plan specified abov | e and agree with its |
| | | Date |
| | | Date |

# **TABLE OF CONTENTS**

| 2.1 Study Objectives 7 2.2 Design Overview 8 Study Duration 12 2.3 Study Treatment 12 2.3.1 Treatment Group 12 2.3.2 Randomization and Blinding 13 2.4 Study Outcome Measures 13 3. SAMPLE SIZE DETERMINATION 13 4. INTERIM ANALYSIS 13 5. ANALYSIS POPULATIONS 13 6. DATA CONVENTION AND RELATED DEFINITIONS 13 6.1 Baseline Definition 14 6.2 Duplicate Data 14 6.3 Handling of Missing Data 14 6.4 Multicenter Clinical Trials 14 6.5 Multiple Comparisons and Type I Error Rate Multiplicity adjustments 14 6.6 Covariates and Prognostic Factors 14 6.7 Stratification Factors 14 6.8 Subgroups and Exploratory Analysis 14 6.9 Standard Calculations 14 6.9.1 Age 14 6.9.2 Weight | Secti | on | | Page |
|---|---|---|---|---|
| 2.1 Study Objectives 7 2.2 Design Overview 8 Study Duration 12 2.3 Study Treatment 12 2.3.1 Treatment Group 12 2.3.2 Randomization and Blinding 13 2.4 Study Outcome Measures 13 3. SAMPLE SIZE DETERMINATION 13 4. INTERIM ANALYSIS 13 5. ANALYSIS POPULATIONS 13 5.1 Safety Population 13 6.1 Baseline Definition 14 6.2 Duplicate Data 14 6.3 Handling of Missing Data 14 6.4 Multicenter Clinical Trials 14 6.5 Multiple Comparisons and Type I Error Rate Multiplicity adjustments 14 6.6 Covariates and Prognostic Factors 14 6.7 Stratification Factors 14 6.8 Subgroups and Exploratory Analysis 14 6.9 Standard Calculations 14 6.9.1 Age 14 6.9.2 Weight 15 < | | LIST | OF ABBREVIATIONS | 5 |
| 2.1 Study Objectives 7 2.2 Design Overview 8 Study Duration 12 2.3 Study Treatment 12 2.3.1 Treatment Group 12 2.3.2 Randomization and Blinding 13 2.4 Study Outcome Measures 13 3. SAMPLE SIZE DETERMINATION 13 4. INTERIM ANALYSIS 13 5.1 Safety Population 13 6.1 Baseline Definition 13 6.1 Baseline Definition 14 6.2 Duplicate Data 14 6.3 Handling of Missing Data 14 6.4 Multicenter Clinical Trials 14 6.5 Multiple Comparisons and Type I Error Rate Multiplicity adjustments 14 6.6 Covariates and Prognostic Factors 14 6.7 Stratification Factors 14 6.8 Subgroups and Exploratory Analysis 14 6.9 Standard Calculations 14 6.9.1 Age 14 6.9.2 Weight 6.6 | 1. | INTR | RODUCTION | 7 |
| 2.2 Design Overview Study Duration 12 | 2. | PRO | PROTOCOL DESIGN AND OBJECTIVES | |
| 2.2 Design Overview Study Duration 12 | | | | |
| Study Duration | | 2.2 | | |
| 2.3 Study Treatment Group 12 2.3.1 Treatment Group 12 2.3.2 Randomization and Blinding 13 2.4 Study Outcome Measures 13 3. SAMPLE SIZE DETERMINATION 13 4. INTERIM ANALYSIS 13 5. ANALYSIS POPULATIONS 13 5.1 Safety Population 13 6. DATA CONVENTION AND RELATED DEFINITIONS 13 6.1 Baseline Definition 14 6.2 Duplicate Data 14 6.3 Handling of Missing Data 14 6.4 Multicenter Clinical Trials 14 6.5 Multiple Comparisons and Type I Error Rate Multiplicity adjustments 14 6.6 Covariates and Prognostic Factors 14 6.7 Stratification Factors 14 6.8 Subgroups and Exploratory Analysis 14 6.9 Standard Calculations 14 6.9.1 Age 14 6.9.2 Weight 15 6.9.3 Change from baseline 15 7.1.1< | | Study | | |
| 2.3.1 Treatment Group | | • | | |
| 2.4 Study Outcome Measures 13 3. SAMPLE SIZE DETERMINATION 13 4. INTERIM ANALYSIS 13 5. ANALYSIS POPULATIONS 13 5.1 Safety Population 13 6. DATA CONVENTION AND RELATED DEFINITIONS 13 6.1 Baseline Definition 14 6.2 Duplicate Data 14 6.3 Handling of Missing Data 14 6.4 Multiple Comparisons and Type I Error Rate Multiplicity adjustments 14 6.5 Multiple Comparisons and Type I Error Rate Multiplicity adjustments 14 6.6 Covariates and Prognostic Factors 14 6.7 Stratification Factors 14 6.8 Subgroups and Exploratory Analysis 14 6.9 Standard Calculations 14 6.9.1 Age 14 6.9.2 Weight 15 6.9.3 Change from baseline 15 7.1 Summarizing and Tabulating the Collected Data 15 7.1.1 Subject Disposition and Withdrawals 15 7.1.2 P | | | 2.3.1 Treatment Group | 12 |
| 3. SAMPLE SIZE DETERMINATION 13 4. INTERIM ANALYSIS 13 5. ANALYSIS POPULATIONS 13 5.1 Safety Population 13 6. DATA CONVENTION AND RELATED DEFINITIONS 13 6.1 Baseline Definition 14 6.2 Duplicate Data 14 6.3 Handling of Missing Data 14 6.4 Multiple Comparisons and Type I Error Rate Multiplicity adjustments 14 6.5 Multiple Comparisons and Type I Error Rate Multiplicity adjustments 14 6.6 Covariates and Prognostic Factors 14 6.7 Stratification Factors 14 6.8 Subgroups and Exploratory Analysis 14 6.9 Standard Calculations 14 6.9.1 Age 14 6.9.2 Weight 15 6.9.3 Change from baseline 15 7.1 SUMMERITY Subject Disposition and Withdrawals 15 7.1.1 Subject Disposition and Withdrawals 15 7.1.2 Protocol Deviations 15 7.1.3 De | | | | |
| 4. INTERIM ANALYSIS 13 5. ANALYSIS POPULATIONS 13 5.1 Safety Population 13 6. DATA CONVENTION AND RELATED DEFINITIONS 13 6.1 Baseline Definition 14 6.2 Duplicate Data 14 6.3 Handling of Missing Data 14 6.4 Multiple Comparisons and Type I Error Rate Multiplicity adjustments 14 6.5 Multiple Comparisons and Type I Error Rate Multiplicity adjustments 14 6.6 Covariates and Prognostic Factors 14 6.7 Stratification Factors 14 6.8 Subgroups and Exploratory Analysis 14 6.9 Standard Calculations 14 6.9.1 Age 14 6.9.2 Weight 15 6.9.3 Change from baseline 15 7.1 Summarizing and Tabulating the Collected Data 15 7.1.1 Subject Disposition and Withdrawals 15 7.1.2 Protocol Deviations 15 7.1.3 Demographics and Baseline Characteristics 16 7.1. | | 2.4 | Study Outcome Measures | 13 |
| 5. ANALYSIS POPULATIONS | 3. | SAM | PLE SIZE DETERMINATION | 13 |
| 5.1 Safety Population 13 6. DATA CONVENTION AND RELATED DEFINITIONS 13 6.1 Baseline Definition 14 6.2 Duplicate Data 14 6.3 Handling of Missing Data 14 6.4 Multicenter Clinical Trials 14 6.5 Multiple Comparisons and Type I Error Rate Multiplicity adjustments 14 6.6 Covariates and Prognostic Factors 14 6.7 Stratification Factors 14 6.8 Subgroups and Exploratory Analysis 14 6.9 Standard Calculations 14 6.9.1 Age 14 6.9.2 Weight 15 6.9.3 Change from baseline 15 7.1 SUMMARIZED 15 7.1 Summarizing and Tabulating the Collected Data 15 7.1.1 Subject Disposition and Withdrawals 15 7.1.2 Protocol Deviations 15 7.1.3 Demographics and Baseline Characteristics 16 7.1.4 Prior and Concomitant Medications 16 7.1.5 Antiretrovir | 4. | INTE | RIM ANALYSIS | 13 |
| 6. DATA CONVENTION AND RELATED DEFINITIONS 13 6.1 Baseline Definition 14 6.2 Duplicate Data 14 6.3 Handling of Missing Data 14 6.4 Multicenter Clinical Trials 14 6.5 Multiple Comparisons and Type I Error Rate Multiplicity adjustments 14 6.6 Covariates and Prognostic Factors 14 6.7 Stratification Factors 14 6.8 Subgroups and Exploratory Analysis 14 6.9 Standard Calculations 14 6.9.1 Age 14 6.9.2 Weight 15 6.9.3 Change from baseline 15 7. STATISTICAL METHODS 15 7.1 Summarizing and Tabulating the Collected Data 15 7.1.1 Subject Disposition and Withdrawals 15 7.1.2 Protocol Deviations 15 7.1.3 Demographics and Baseline Characteristics 16 7.1.4 Prior and Concomitant Medications 16 7.1.5 Antiretroviral Therapy 16 7.1.6 < | 5. | ANA | LYSIS POPULATIONS | 13 |
| 6.1 Baseline Definition 14 6.2 Duplicate Data 14 6.3 Handling of Missing Data 14 6.4 Multicenter Clinical Trials 14 6.5 Multiple Comparisons and Type I Error Rate Multiplicity adjustments 14 6.6 Covariates and Prognostic Factors 14 6.7 Stratification Factors 14 6.8 Subgroups and Exploratory Analysis 14 6.9 Standard Calculations 14 6.9.1 Age 14 6.9.2 Weight 15 6.9.3 Change from baseline 15 7.1 Summarizing and Tabulating the Collected Data 15 7.1.1 Subject Disposition and Withdrawals 15 7.1.2 Protocol Deviations 15 7.1.2 Protocol Deviations 15 7.1.3 Demographics and Baseline Characteristics 16 7.1.4 Prior and Concomitant Medications 16 7.1.5 Antiretroviral Therapy 16 7.1.6 Optimized Background Therapy (OBT) 16 7.1.7 | | 5.1 | Safety Population | 13 |
| 6.2 Duplicate Data 14 6.3 Handling of Missing Data. 14 6.4 Multicenter Clinical Trials 14 6.5 Multiple Comparisons and Type I Error Rate Multiplicity adjustments 14 6.6 Covariates and Prognostic Factors 14 6.7 Stratification Factors 14 6.8 Subgroups and Exploratory Analysis 14 6.9 Standard Calculations 14 6.9.1 Age 14 6.9.2 Weight 15 6.9.3 Change from baseline 15 7.1 Summarizing and Tabulating the Collected Data 15 7.1.1 Subject Disposition and Withdrawals 15 7.1.2 Protocol Deviations 15 7.1.2 Protocol Deviations 15 7.1.3 Demographics and Baseline Characteristics 16 7.1.4 Prior and Concomitant Medications 16 7.1.5 Antiretroviral Therapy 16 6.7.1.7 Treatment Administration 17 7.2 Analysis of Study Outcome Measures 17 7.2.1 <td>6.</td> <td>DAT</td> <td>A CONVENTION AND RELATED DEFINITIONS</td> <td>13</td> | 6. | DAT | A CONVENTION AND RELATED DEFINITIONS | 13 |
| 6.2 Duplicate Data 14 6.3 Handling of Missing Data. 14 6.4 Multicenter Clinical Trials 14 6.5 Multiple Comparisons and Type I Error Rate Multiplicity adjustments 14 6.6 Covariates and Prognostic Factors 14 6.7 Stratification Factors 14 6.8 Subgroups and Exploratory Analysis 14 6.9 Standard Calculations 14 6.9.1 Age 14 6.9.2 Weight 15 6.9.3 Change from baseline 15 7.1 Summarizing and Tabulating the Collected Data 15 7.1.1 Subject Disposition and Withdrawals 15 7.1.2 Protocol Deviations 15 7.1.2 Protocol Deviations 15 7.1.3 Demographics and Baseline Characteristics 16 7.1.4 Prior and Concomitant Medications 16 7.1.5 Antiretroviral Therapy 16 6.7.1.7 Treatment Administration 17 7.2 Analysis of Study Outcome Measures 17 7.2.1 <td></td> <td>6.1</td> <td>Baseline Definition</td> <td>14</td> | | 6.1 | Baseline Definition | 14 |
| 6.3 Handling of Missing Data. 14 6.4 Multiple Comparisons and Type I Error Rate Multiplicity adjustments. 14 6.5 Multiple Comparisons and Type I Error Rate Multiplicity adjustments. 14 6.6 Covariates and Prognostic Factors. 14 6.7 Stratification Factors. 14 6.8 Subgroups and Exploratory Analysis. 14 6.9 Standard Calculations. 14 6.9.1 Age. 14 6.9.2 Weight. 15 6.9.3 Change from baseline. 15 7.1 Summarizing and Tabulating the Collected Data 15 7.1.1 Subject Disposition and Withdrawals 15 7.1.2 Protocol Deviations 15 7.1.2 Protocol Deviations 15 7.1.3 Demographics and Baseline Characteristics 16 7.1.4 Prior and Concomitant Medications 16 7.1.5 Antiretroviral Therapy 16 7.1.6 Optimized Background Therapy (OBT) 16 7.1.7 Treatment Administration 17 7.2.1 Mean change in viral load | | 6.2 | | |
| 6.4 Multicenter Clinical Trials 14 6.5 Multiple Comparisons and Type I Error Rate Multiplicity adjustments 14 6.6 Covariates and Prognostic Factors 14 6.7 Stratification Factors 14 6.8 Subgroups and Exploratory Analysis 14 6.9 Standard Calculations 14 6.9.1 Age 14 6.9.2 Weight 15 6.9.3 Change from baseline 15 7. STATISTICAL METHODS 15 7.1 Summarizing and Tabulating the Collected Data 15 7.1.1 Subject Disposition and Withdrawals 15 7.1.2 Protocol Deviations 15 7.1.3 Demographics and Baseline Characteristics 16 7.1.4 Prior and Concomitant Medications 16 7.1.5 Antiretroviral Therapy 16 7.1.6 Optimized Background Therapy (OBT) 16 7.1.7 Treatment Administration 17 7.2 Analysis of Study Outcome Measures 17 7.2.1 Mean change in viral load (HIV-1 RNA levels) 17 | | 6.3 | 1 | |
| 6.6 Covariates and Prognostic Factors 14 6.7 Stratification Factors 14 6.8 Subgroups and Exploratory Analysis 14 6.9 Standard Calculations 14 6.9.1 Age 14 6.9.2 Weight 15 6.9.3 Change from baseline 15 7.1 Summarizing and Tabulating the Collected Data 15 7.1.1 Subject Disposition and Withdrawals 15 7.1.2 Protocol Deviations 15 7.1.3 Demographics and Baseline Characteristics 16 7.1.4 Prior and Concomitant Medications 16 7.1.5 Antiretroviral Therapy 16 7.1.6 Optimized Background Therapy (OBT) 16 7.1.7 Treatment Administration 17 7.2 Analysis of Study Outcome Measures 17 7.2.1 Mean change in viral load (HIV-1 RNA levels) 17 7.2.2 Mean change in inviral load (MIV-1 RNA levels) 17 7.2.3 Emergence of Dual/Mixed (D/M) - and CXCR4-tropic virus 18 7.2.4 Analysis of Safety Data | | 6.4 | | |
| 6.7 Stratification Factors 14 6.8 Subgroups and Exploratory Analysis 14 6.9 Standard Calculations 14 6.9.1 Age 14 6.9.2 Weight 15 6.9.3 Change from baseline 15 7.1 Summarizing and Tabulating the Collected Data 15 7.1.1 Subject Disposition and Withdrawals 15 7.1.2 Protocol Deviations 15 7.1.3 Demographics and Baseline Characteristics 16 7.1.4 Prior and Concomitant Medications 16 7.1.5 Antiretroviral Therapy 16 7.1.6 Optimized Background Therapy (OBT) 16 7.1.7 Treatment Administration 17 7.2 Analysis of Study Outcome Measures 17 7.2.1 Mean change in viral load (HIV-1 RNA levels) 17 7.2.2 Mean change in in CD4 cell count 17 7.2.3 Emergence of Dual/Mixed (D/M) - and CXCR4-tropic virus 18 7.2.4 Analysis of Safety Data 18 7.2.5 Clinical Laboratory Evaluations 19 <td></td> <td>6.5</td> <td>Multiple Comparisons and Type I Error Rate Multiplicity adjustments</td> <td>14</td> | | 6.5 | Multiple Comparisons and Type I Error Rate Multiplicity adjustments | 14 |
| 6.8 Subgroups and Exploratory Analysis 14 6.9 Standard Calculations 14 6.9.1 Age 14 6.9.2 Weight 15 6.9.3 Change from baseline 15 7. STATISTICAL METHODS 15 7.1 Summarizing and Tabulating the Collected Data 15 7.1.1 Subject Disposition and Withdrawals 15 7.1.2 Protocol Deviations 15 7.1.3 Demographics and Baseline Characteristics 16 7.1.4 Prior and Concomitant Medications 16 7.1.5 Antiretroviral Therapy 16 7.1.6 Optimized Background Therapy (OBT) 16 7.1.7 Treatment Administration 17 7.2 Analysis of Study Outcome Measures 17 7.2.1 Mean change in viral load (HIV-1 RNA levels) 17 7.2.2 Mean change in CD4 cell count 17 7.2.3 Emergence of Dual/Mixed (D/M) - and CXCR4-tropic virus 18 7.2.4 Analysis of Safety Data 18 7.2.5 Clinical Laboratory Evaluations 19 | | 6.6 | Covariates and Prognostic Factors | 14 |
| 6.9 Standard Calculations 14 6.9.1 Age 14 6.9.2 Weight 15 6.9.3 Change from baseline 15 7. STATISTICAL METHODS 15 7.1 Summarizing and Tabulating the Collected Data 15 7.1.1 Subject Disposition and Withdrawals 15 7.1.2 Protocol Deviations 15 7.1.3 Demographics and Baseline Characteristics 16 7.1.4 Prior and Concomitant Medications 16 7.1.5 Antiretroviral Therapy 16 7.1.6 Optimized Background Therapy (OBT) 16 7.1.7 Treatment Administration 17 7.2 Analysis of Study Outcome Measures 17 7.2.1 Mean change in viral load (HIV-1 RNA levels) 17 7.2.2 Mean change in CD4 cell count 17 7.2.3 Emergence of Dual/Mixed (D/M) - and CXCR4-tropic virus 18 7.2.4 Analysis of Safety Data 18 7.2.5 Clinical Laboratory Evaluations 19 | | 6.7 | Stratification Factors | 14 |
| 6.9.1 Age 14 6.9.2 Weight 15 6.9.3 Change from baseline 15 7. STATISTICAL METHODS 15 7.1 Summarizing and Tabulating the Collected Data 15 7.1.1 Subject Disposition and Withdrawals 15 7.1.2 Protocol Deviations 15 7.1.3 Demographics and Baseline Characteristics 16 7.1.4 Prior and Concomitant Medications 16 7.1.5 Antiretroviral Therapy 16 7.1.6 Optimized Background Therapy (OBT) 16 7.1.7 Treatment Administration 17 7.2 Analysis of Study Outcome Measures 17 7.2.1 Mean change in viral load (HIV-1 RNA levels) 17 7.2.2 Mean change in CD4 cell count 17 7.2.3 Emergence of Dual/Mixed (D/M) - and CXCR4-tropic virus 18 7.2.4 Analysis of Safety Data 18 7.2.5 Clinical Laboratory Evaluations 19 | | 6.8 | Subgroups and Exploratory Analysis | 14 |
| 6.9.2 Weight. 15 6.9.3 Change from baseline 15 7. STATISTICAL METHODS. 15 7.1 Summarizing and Tabulating the Collected Data 15 7.1.1 Subject Disposition and Withdrawals 15 7.1.2 Protocol Deviations 15 7.1.3 Demographics and Baseline Characteristics 16 7.1.4 Prior and Concomitant Medications 16 7.1.5 Antiretroviral Therapy 16 7.1.6 Optimized Background Therapy (OBT) 16 7.1.7 Treatment Administration 17 7.2 Analysis of Study Outcome Measures 17 7.2.1 Mean change in viral load (HIV-1 RNA levels) 17 7.2.2 Mean change in CD4 cell count 17 7.2.3 Emergence of Dual/Mixed (D/M) - and CXCR4-tropic virus 18 7.2.4 Analysis of Safety Data 18 7.2.5 Clinical Laboratory Evaluations 19 | | 6.9 | Standard Calculations | 14 |
| 6.9.3 Change from baseline 15 7. STATISTICAL METHODS | | | | |
| 7. STATISTICAL METHODS | | | | |
| 7.1 Summarizing and Tabulating the Collected Data 15 7.1.1 Subject Disposition and Withdrawals 15 7.1.2 Protocol Deviations 15 7.1.3 Demographics and Baseline Characteristics 16 7.1.4 Prior and Concomitant Medications 16 7.1.5 Antiretroviral Therapy 16 7.1.6 Optimized Background Therapy (OBT) 16 7.1.7 Treatment Administration 17 7.2 Analysis of Study Outcome Measures 17 7.2.1 Mean change in viral load (HIV-1 RNA levels) 17 7.2.2 Mean change in CD4 cell count 17 7.2.3 Emergence of Dual/Mixed (D/M) - and CXCR4-tropic virus 18 7.2.4 Analysis of Safety Data 18 7.2.5 Clinical Laboratory Evaluations 19 | _ | | | |
| 7.1.1 Subject Disposition and Withdrawals 15 7.1.2 Protocol Deviations 15 7.1.3 Demographics and Baseline Characteristics 16 7.1.4 Prior and Concomitant Medications 16 7.1.5 Antiretroviral Therapy 16 7.1.6 Optimized Background Therapy (OBT) 16 7.1.7 Treatment Administration 17 7.2 Analysis of Study Outcome Measures 17 7.2.1 Mean change in viral load (HIV-1 RNA levels) 17 7.2.2 Mean change in CD4 cell count 17 7.2.3 Emergence of Dual/Mixed (D/M) - and CXCR4-tropic virus 18 7.2.4 Analysis of Safety Data 18 7.2.5 Clinical Laboratory Evaluations 19 | 7. | | | |
| 7.1.2 Protocol Deviations 15 7.1.3 Demographics and Baseline Characteristics 16 7.1.4 Prior and Concomitant Medications 16 7.1.5 Antiretroviral Therapy 16 7.1.6 Optimized Background Therapy (OBT) 16 7.1.7 Treatment Administration 17 7.2 Analysis of Study Outcome Measures 17 7.2.1 Mean change in viral load (HIV-1 RNA levels) 17 7.2.2 Mean change in CD4 cell count 17 7.2.3 Emergence of Dual/Mixed (D/M) - and CXCR4-tropic virus 18 7.2.4 Analysis of Safety Data 18 7.2.5 Clinical Laboratory Evaluations 19 | | 7.1 | | |
| 7.1.3 Demographics and Baseline Characteristics 16 7.1.4 Prior and Concomitant Medications 16 7.1.5 Antiretroviral Therapy 16 7.1.6 Optimized Background Therapy (OBT) 16 7.1.7 Treatment Administration 17 7.2 Analysis of Study Outcome Measures 17 7.2.1 Mean change in viral load (HIV-1 RNA levels) 17 7.2.2 Mean change in CD4 cell count 17 7.2.3 Emergence of Dual/Mixed (D/M) - and CXCR4-tropic virus 18 7.2.4 Analysis of Safety Data 18 7.2.5 Clinical Laboratory Evaluations 19 | | | | |
| 7.1.4 Prior and Concomitant Medications 16 7.1.5 Antiretroviral Therapy 16 7.1.6 Optimized Background Therapy (OBT) 16 7.1.7 Treatment Administration 17 7.2 Analysis of Study Outcome Measures 17 7.2.1 Mean change in viral load (HIV-1 RNA levels) 17 7.2.2 Mean change in CD4 cell count 17 7.2.3 Emergence of Dual/Mixed (D/M) - and CXCR4-tropic virus 18 7.2.4 Analysis of Safety Data 18 7.2.5 Clinical Laboratory Evaluations 19 | | | | |
| 7.1.5 Antiretroviral Therapy 16 7.1.6 Optimized Background Therapy (OBT) 16 7.1.7 Treatment Administration 17 7.2 Analysis of Study Outcome Measures 17 7.2.1 Mean change in viral load (HIV-1 RNA levels) 17 7.2.2 Mean change in CD4 cell count 17 7.2.3 Emergence of Dual/Mixed (D/M) - and CXCR4-tropic virus 18 7.2.4 Analysis of Safety Data 18 7.2.5 Clinical Laboratory Evaluations 19 | | | C 1 | |
| 7.1.6 Optimized Background Therapy (OBT) 16 7.1.7 Treatment Administration 17 7.2 Analysis of Study Outcome Measures 17 7.2.1 Mean change in viral load (HIV-1 RNA levels) 17 7.2.2 Mean change in CD4 cell count 17 7.2.3 Emergence of Dual/Mixed (D/M) - and CXCR4-tropic virus 18 7.2.4 Analysis of Safety Data 18 7.2.5 Clinical Laboratory Evaluations 19 | | | | |
| 7.2Analysis of Study Outcome Measures177.2.1Mean change in viral load (HIV-1 RNA levels)177.2.2Mean change in CD4 cell count177.2.3Emergence of Dual/Mixed (D/M) - and CXCR4-tropic virus187.2.4Analysis of Safety Data187.2.5Clinical Laboratory Evaluations19 | | | 7.1.6 Optimized Background Therapy (OBT) | 16 |
| 7.2.1 Mean change in viral load (HIV-1 RNA levels) 17 7.2.2 Mean change in CD4 cell count 17 7.2.3 Emergence of Dual/Mixed (D/M) - and CXCR4-tropic virus 18 7.2.4 Analysis of Safety Data 18 7.2.5 Clinical Laboratory Evaluations 19 | | | 7.1.7 Treatment Administration | 17 |
| 7.2.2 Mean change in CD4 cell count 17 7.2.3 Emergence of Dual/Mixed (D/M) - and CXCR4-tropic virus 18 7.2.4 Analysis of Safety Data 18 7.2.5 Clinical Laboratory Evaluations 19 | | 7.2 | | |
| 7.2.3 Emergence of Dual/Mixed (D/M) - and CXCR4-tropic virus 18 7.2.4 Analysis of Safety Data 18 7.2.5 Clinical Laboratory Evaluations 19 | | | · | |
| 7.2.4 Analysis of Safety Data | | | 6 | |
| 7.2.5 Clinical Laboratory Evaluations | | | | |

| -, | J | | | - **** |
|---|---|---|---|---|
| | | 7.2.8 | Vital Signs Electrocardiogram (ECGs) | 19 |
| 8. | A DDI | | Additional Data listings and tabulations SCHEDULE OF ASSESSMENTS | |
| 9. | APPI | | - PLANNED TLG | |
| | 9.1 | Planne | d by-subject listings | 24 |
| | 9.2 | Planne | d Summary Tables | 25 |
| 11. | VER | SION HIS | STORY | 27 |

# LIST OF ABBREVIATIONS

| Abbreviation | Term |
|--------------|----------------------------------------------|
| AE | Adverse Event |
| ALT | Alanine Transaminase |
| ANC | Absolute Neutrophil Count |
| ART | Anti Retroviral Therapy |
| AST | Aspartate Transaminase |
| ATC | Anatomic Therapeutic Classification |
| CBC | Complete Blood Count |
| CCR5 | C-C chemokine receptor type 5 |
| CS | Clinically Significant |
| DAIDS | Division of AIDS |
| DNA | Deoxyribonucleic Acid |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| et al | et aliae; Latin for "and others" |
| EOT | End of Treatment |
| EOT2 | End of Treatment Extension |
| °F | Fahrenheit |
| FU | Follow-Up |
| HAART | Highly Active Antiretroviral Therapy |
| HBsAg | Hepatitis B Surface Antigen |
| HCT | Hematocrit |
| HIV | Human Immunodeficiency Virus |
| ICH | International Conference on Harmonization |
| i.e. | id est; Latin for "that is" |
| INR | International Normalized Ratio |
| IP | Investigational Product |
| ISR | Injection Site Reactions |
| LAR | Legally Acceptable Representative |
| LDH | Lactate dehydrogenase |
| LPN | Licensed Practical Nurse |
| LVN | Licensed Vocational Nurse |
| MD | Doctor of Medicine |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram |
| mL | Milliliter |
| Abbreviation | Term |

| mm | Millimeter |
|------|-----------------------------------|
| NCS | Not Clinically Significant |
| NP | Nurse Practitioner |
| NVF | Non-Virologic Failure |
| OBT | Optimized Background Therapy |
| PA | Physician Assistant |
| PI | Principal Investigator |
| PK | Pharmacokinetics |
| PP | Per Protocol |
| RBC | Red Blood Cells |
| RN | Registered Nurse |
| RNA | Ribonucleic acid |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SC | Subcutaneous |
| SD | Standard Deviation |
| TE | Treatment Extension |
| TEAE | Treatment Emergent Adverse Events |
| VF | Virologic Failure |
| WBC | White Blood Cells |

#### 1. INTRODUCTION

This Statistical Analysis Plan describes the planned analyses and reporting for the clinical trial protocol PRO 140\_CD01-Extension, sponsored by CytoDyn Inc. The reader of this Statistical Analysis Plan (SAP) is encouraged to review the complete protocol and amendments as this plan contains only a limited overview of protocol information. The main objective of this plan is to provide details pertaining to statistical methodology, data conventions, and processes used for the analysis of data from this trial.

The format and content of this Statistical Analysis Plan are structured to provide sufficient detail to meet the requirements specified by the International Conference on Harmonization (ICH) E9: Guidance on Statistical Principles in Clinical Trials. All work planned and presented in this Statistical Analysis Plan will follow the ethical guidelines published by the American Statistical Association (ASA).

The following documents were reviewed in preparation of this Statistical Analysis Plan:

- Version 4.0, protocol 13 May 2019
- ASA Ethical Guidelines for Statistical Practice (2016)
- The Royal Statistical Society: Code of Conduct (2014)
- ICH Guidance on the Structure and Content of Clinical Study Reports (ICH E3, 1996)
- ICH Guidance on the Structure and Content of Clinical Study Reports (ICH E3(R1), 2013)
- ICH Guidance on the Statistical Principles for Clinical Trials (ICH E9, 1998)
- ICH Guidance on the Statistical Principles for Clinical Trials (ICH E9(R1), 2017)

#### 2. PROTOCOL DESIGN AND OBJECTIVES

#### 2.1 Study Objectives

The primary objective is to provide PRO 140 on a continued basis to subjects who complete participation in PRO140\_CD02 or CD02\_OpenLabel and would require continued access to PRO 140 to form a viable regimen, in the opinion of the treating physician.

**Study Center:** Up to 10 centers in the United States. Centers must have the capability of implementing appropriate infection-control measures to prevent infection of study staff and others who share the clinical site space.

#### 2.2 Design Overview

This is an extension study, to provide continued access to PRO 140 to subjects who complete participation in PRO140\_CD02 or CD02\_OpenLabel and continue to receive clinical benefit and would require PRO 140 to form a viable regimen, in the opinion of the treating physician. The patient population for this trial is treatment-experienced HIV-infected patients with CCR5-tropic virus who demonstrate evidence of HIV-1 suppression after successfully completed 24 weeks of treatment in the PRO140 CD02 or CD02 Open Label study.

PRO 140 700 mg is administered as subcutaneous injection in the abdomen weekly. A total of 700 mg (175 mg/mL) is delivered as two 2 mL injections on opposite sides of the abdomen. Subjects who were enrolled under a previous Protocol version and are still receiving the 350 mg dose, have the option of increasing their dose to 700mg for the remainder of the Treatment Extension Phase to provide maximum viral load suppression in a heavily treatment experienced population to avoid developing resistance to current OBT therapies.

**NOTE:** Alternatively, the 700 mg dose may be delivered as four 1mL doses (two SC injections on opposite sides of abdomen) for those that experience discomfort with the 2mL injections (i.e. subjects with low body fat percentages).

The study will have three phases: Screening Phase, Treatment Extension Phase and Follow-up Phase as shown in the study flow diagram **Figure 2-1**.

#### **Screening Phase (up to 21days):**

This phase is designed to determine whether subjects are eligible to proceed to the Treatment Phase of the study. This phase consists of a series of assessments designed to determine eligibility. A written informed consent from the subject will be obtained by the Investigator or suitably qualified individual before the performance of any protocol-specific procedure.

All subjects will continue taking PRO 140 along with OBT during the Screening Phase.

**NOTE:** Subject consent and screening assessments should be completed prior to EOT visit in the PRO140\_CD02 or CD02\_OpenLabel study.

### **Treatment Extension Phase:**

The Treatment Extension Phase begins with an evaluation of most recent laboratory results (viral load & CD4 count) obtained in PRO140\_CD02 or CD02\_OpenLabel study. All subjects who fail to meet eligibility criteria will be considered screen failures and exit the study without further evaluation. Subjects who meet all eligibility criteria will receive first treatment injection at Treatment Extension (TE) Visit 1 (which corresponds to EOT from PRO140\_CD02 or CD02\_OpenLabel study).

The Treatment Extension Phase consists of weekly treatment injections of PRO140 700mg\* SC in addition to OBT. Optimized background therapy (OBT) is a standard-of-care regimen comprised of 3 or more antiretroviral agents selected by the Investigator based on treatment history and genotypic and/or phenotypic assessments. Subjects will continue the same OBT regimen initiated within the PRO140 CD02 or CD02 OpenLabel study.

**NOTE:** Subjects enrolled prior to Protocol v4.0 may still be receiving the original 350mg dose and have the option of increasing their dose to 700mg.

As shown in Table 0-1, all subjects will receive PRO 140 SC injection and Optimized Background Therapy.

The injectable study treatment (PRO 140) will be administered:

- by a qualified medical professional (MD, DO, PA, LPN, LVN, NP, RN, or CMA if permitted by state law) or
- self-administered by subjects

Study participants will be monitored every 4 weeks for viral load and CD4 count. Should subjects experience virologic failure, they will be allowed to continue PRO 140 with existing OBT regimen while waiting for new regimen to be constructed by the Investigator.

Virologic failure is defined two consecutive HIV-1 RNA levels  $\geq$  400 copies/mL.

Subjects who experience virologic failure at any point during the Treatment Extension Phase will undergo the Virologic Failure (VF) Visit assessments and then return in 4 weeks ( $\pm$  allowed window) for the Safety Follow-up Visits.

# **Safety Follow-up Visit:**

Duration of the Follow-up Phase is determined upon whether or not subject has experienced virologic failure during the Treatment Extension Phase.

- Subjects who experience virologic failure within Treatment Extension Phase will be followed up every 4 weeks until viral suppression is achieved (i.e., plasma HIV-1 RNA levels below level of detection) or up to a maximum of 6 months after cessation of therapy if the treating physician does not feel that there is an antiretroviral regimen that will regain full viral suppression.
- Subjects who do not experience virologic failure at the end of Treatment Extension Phase, will be followed up every 2 weeks for total of 4 weeks.



Figure 2-1 Clinical Trial Flow Diagram

#### **Study Duration**

# Screening Phase:

o up to 21 days

#### • Treatment Extension Phase:

 weekly (± allowed windows) until subject withdraws consent, experience virologic failure or PRO 140 is approved or CytoDyn decides to discontinue its development

#### Follow-up Phase:

weeks\* (± allowed windows)

\*or up to maximum of 6 months after experiencing Virologic Failure (VF) if the treating physician does not feel that there is an antiretroviral regimen that will regain full viral suppression.

#### 2.3 Study Treatment

### 2.3.1 Treatment Group

This is a single arm study. All eligible subjects will receive PRO 140 SC injection and Optimized Background Therapy. PRO 140 as a 350mg dose (per protocol prior to v4.0) or 700mg (per protocol after v4.0) subcutaneous injection weekly until one of the following occurs:

- Virologic failure
- Consent withdrawn
- PRO 140 is approved
- CytoDyn decides to discontinue its development

**NOTE:** Subjects enrolled prior to Protocol v4.0 may still be receiving the original 350mg dose and have the option of increasing their dose to 700mg.

| Study Drug | Dosage Form | IP<br>concentration | Dosing Frequency and<br>Amount | Route of<br>Administration |
|---|---|---|---|---|
| | | | 2 injections of PRO 140<br>(2 X 1 mL/inj.) | |
| | Parenteral | | for 48 weeks | |
| PRO 140 350mg | solution | 175 mg/mL | for 48 weeks | SC injection |

| DD 0 140 700 | Parenteral | 175 /I | 2 injections of PRO 140<br>(2 X 2 mL/inj.) | SC initiation | |
|---|---|---|---|---|---|
| PRO 140 700mg | solution | 175 mg/mL | for 48 weeks | SC injection | ı |

# 2.3.2 Randomization and Blinding

No blinding or randomization requirement.

#### 2.4 Study Outcome Measures

- Mean change in viral load (HIV-1 RNA levels) at the conclusion of treatment period
- Mean change in CD4 cell count at the conclusion of treatment period
- Emergence of Dual/Mixed (D/M)- and CXCR4-tropic virus in patients who had exclusive CCR5-tropic virus at study entry.
- Tolerability of repeated subcutaneous administration of PRO 140 as assessed by investigatorevaluation of injection site reactions
- Frequency of treatment-related adverse events resulting in study drug discontinuation
- Frequency of Grade 3 or 4 adverse events as defined by the DAIDS Adverse Event scale

#### 3. SAMPLE SIZE DETERMINATION

Sample size determination is not applicable as only those subjects who are currently enrolled in PRO 140\_CD 02 or CD02\_OpenLabel study are allowed to participate in this study.

#### 4. INTERIM ANALYSIS

There is no planned interim analysis (IA) for this study.

#### 5. ANALYSIS POPULATIONS

## 5.1 Safety Population

The Safety population is defined as the set of subjects who received at least one dose of PRO 140. This population will be used for the analysis of safety parameters.

#### 6. DATA CONVENTION AND RELATED DEFINITIONS

#### 6.1 Baseline Definition

Baseline for a given parameter or endpoint is defined to be the baseline of CD02 or CD02\_OpenLabel study.

### 6.2 Duplicate Data

For unplanned duplicate data within a protocol-specified visit, the last measured value will be used for the analysis. If it is not possible to identify the "last measured value" the average of the duplicate values will be used.

#### 6.3 Handling of Missing Data

There will be no imputation of missing data for this study.

#### 6.4 Multicenter Clinical Trials

Up to 30 centers in the United States.

#### 6.5 Multiple Comparisons and Type I Error Rate Multiplicity adjustments

This is a proof of concept study and there is no need for adjustment of Type I error rate.

# 6.6 Covariates and Prognostic Factors

There are no pre-planned covariates analyses of the data from this study.

#### 6.7 Stratification Factors

There are no stratification factors for this study.

#### 6.8 Subgroups and Exploratory Analysis

There are no subgroups and exploratory analysis for this study.

#### 6.9 Standard Calculations

#### 6.9.1 Age

Age will be calculated as the number of completed years between the date of informed consent and the subject's birth date.

Age (years) = integer of [(date of informed consent - date of birth)/365.25 + 0.5]

### 6.9.2 Weight

For summary purposes weight will be expressed in kilograms. Entries made in pounds will be converted to kilograms using the formula noted below.

Weight (kg) = Weight (lb)/
$$2.2046$$

# 6.9.3 Change from baseline

Change from baseline will be calculated for each post baseline visit as follows:

Change From Baseline = Post baseline result at time t - Baseline result

#### 7. STATISTICAL METHODS

All collected study data will be presented in subject data listings. Statistical analyses will be performed using SAS® for Windows, version 9.4 or later.

## 7.1 Summarizing and Tabulating the Collected Data

All data collected will be summarized according to the variable type:

- Continuous data summaries will include number of observations, mean, standard deviation, median, and minimum and maximum values.
- Categorical data summaries will include frequency counts and percentages.

#### 7.1.1 Subject Disposition and Withdrawals

- There will be a detailed accounting of all subjects that signed the informed consent to
  participate in this trial. The following will be summarized: The number of subjects who are
  screenedThe number of subjects who received treatment
- The number of subjects who completed the study
- The number of subjects who discontinued during the study
- The reason for all post treatment study discontinuation

In addition, there will also be a listing of all discontinued subjects, which will provide the specific reason for discontinuation.

#### 7.1.2 Protocol Deviations

The deviations occurring during the clinical trial will be summarized descriptively according to the following categories:

- Informed Consent deviation
- Inclusion/Exclusion criteria deviation
- Developed withdrawal criteria deviation
- Procedure performed out of window
- Received an excluded concomitant medication
- Missed procedure
- All other deviations

Additionally a by-subject listing of all deviations will also be prepared.

#### 7.1.3 Demographics and Baseline Characteristics

Demographic and baseline characteristics (i.e., Age, Gender, Time since HIV diagnosis, Viral load at T1, etc.) will be summarized using appropriate descriptive statistics.

Medical history of the subjects will also be provided as a by-subject listing.

#### 7.1.4 Prior and Concomitant Medications

Prior and concomitant medications will be summarized for the Safety population. All prior and concomitant medications recorded in the eCRFs will be coded to generic term and all matching Anatomic Therapeutic Classification (ATC) codes using WHO Drug Summaries will be prepared using the coded terms. All prior and concomitant medications recorded in the eCRFs will also be listed.

#### 7.1.5 Antiretroviral Therapy

Antiretroviral Therapy is not captured in this study but data captured in the PRO140\_CD02 and PR140\_CD02 Open Label used to summarize the data for to PRO140\_CD02\_Extension.

Anti-retroviral therapy will be summarized for the Safety Population. All such medications recorded in the eCRFs will be coded to generic term and all matching Anatomic Therapeutic Classification (ATC) codes using WHO Drug. Summaries will be prepared using the coded terms. All anti-retroviral therapy recorded in the eCRFs will also be listed.

# 7.1.6 Optimized Background Therapy (OBT)

Optimized background therapy will be summarized for the Safety Population. All such medications recorded in the eCRFs will be coded to generic term and all matching Anatomic Therapeutic

Classification (ATC) codes using WHO Drug. Summaries will be prepared using the coded terms. All optimized background therapy recorded in the eCRFs will also be listed.

#### 7.1.7 Treatment Administration

PRO 140 will be administered as a 350mg subcutaneous injection weekly during treatment extension phase in addition to OBT.

A total of 700 mg (175 mg/mL) is delivered as two 2 mL injections administered subcutaneously on opposite sides of the abdomen.

Subjects who were enrolled under a Protocol version 4.0 and are still receiving the 350 mg dose, have the option of increasing their dose to 700mg for the remainder of the Treatment Extension Phase.

**Note**: IP must be administered by a qualified medical professional (MD, DO, PA, LPN, LVN, NP, RN or CMA if permitted by state law) or self-administered by subjects.

All treatment PRO-140 administration data will be listed. In addition, the number and percentage of the subjects who received PRO-140 injection will be presented for the safety population for each week during the treatment period.

### 7.2 Analysis of Study Outcome Measures

The analysis of study outcome measure will be conducted on the safety population.

## 7.2.1 Mean change in viral load (HIV-1 RNA levels)

The raw and change from baseline in HIV-1 RNA levels (log10 copies/mL) will be summarized atleast once every four week during the treatment extension phase. For change from baseline summaries, subjects with an undefined change from baseline, because of missing data, will be excluded.

# 7.2.2 Mean change in CD4 cell count

The raw and change from baseline in CD4 cell count will be summarized for each week during the treatment phase. The summary tables will include the number of observations, mean, standard deviation, median, and minimum and maximum values. For change from baseline summaries, subjects with an undefined change from baseline, because of missing data, will be excluded.

# 7.2.3 Emergence of Dual/Mixed (D/M) - and CXCR4-tropic virus

The data for this outcome measure will be provided by external vendor Monogram Biosciences. All patients have exclusive CCR5-tropic (i.e., R5 or X4) virus at study entry. The proportion of subjects with any tropism result of dual/mixed will be summarized.

# 7.2.4 Analysis of Safety Data

The Safety population will be used for the analysis of safety endpoints. No inferential statistics are planned.

#### 7.2.4.1 Adverse Events

Adverse events will be classified by system organ class and preferred term (PT) according to the most recent MedDRA dictionary.

Since this is an extension of the PRO 140\_CD 02 study, all adverse events (AE) that captured in this study will be considered as Treatment Emergent Adverse Events (TEAEs). The following TEAE summaries will be provided, using frequency counts and percentages:

- Overall (*i.e.*, regardless of severity or relationship to treatment)
- By severity grade (mild, moderate, severe, life threatening or death)
- By relationship to study treatment

In addition, separate summaries of SAEs, and AEs resulting in discontinuation of study treatment will be presented.

Unless otherwise specified, at each level of subject summarization, a subject will be counted only once. If there is more than one occurrence of an event, the event of the worst severity or the worst-case relationship category will be summarized.

#### 7.2.4.2 Tolerability Assessment

#### 7.2.4.3 Injection Site Reaction

At each visit during the Treatment Extension Phase, an injection site reaction assessment will be made for the current and previous injection sites. Injection site reaction assessments are recorded by the Investigator starting after the first injection is given. All data from the injection site reaction assessments of the repeated subcutaneous administration of PRO 140 will be presented and descriptively summarized.

### 7.2.5 Clinical Laboratory Evaluations

All available results of the clinical laboratory evaluations will be listed and summarized. Laboratory evaluations include hematology (routine CBC), biochemistry, coagulation indices, urinalysis, glomerular filtration rate (GFR) and HBsAg etc.

#### 7.2.5.1 Laboratory Values over Time

Summary statistics of raw data and change from baseline values for each laboratory parameter will be presented. Data will be summarized as appropriate to the variable type.

For change from baseline summaries, subjects with an undefined change from baseline, because of missing data, will be excluded.

#### 7.2.5.2 Individual Subject Changes (Shift Tables)

Individual subject changes will be identified through shift tables. Shift tables will be presented for each laboratory parameter with counts and percentages of subjects, for shift (change) from baseline.

#### 7.2.6 Physical Examination

All physical examination findings will be listed and/or summarized.

# 7.2.7 Vital Signs

Tabulations of raw data and change from baseline values will be presented by time point for each vital sign parameter [*i.e.*, Heart Rate (beats/min), temperature ( ${}^{0}C / {}^{0}F$ ), systolic BP (mmHg), diastolic BP (mmHg), and Respiration Rate].

Tabulations will include the number of observations, mean, standard deviation, median, and minimum and maximum values. For change from baseline summaries, subjects with an undefined change from baseline, because of missing data, will be excluded.

# 7.2.8 Electrocardiogram (ECGs)

All ECGs findings will be listed and/or summarized. The following parameters will be recorded: ventricular rate (beats per minute), PR interval (msec), QRS interval (msec), QT interval (msec), and QTc interval (msec). Additionally, the investigator will record the overall results of the ECG reading as either normal or abnormal, and as either not clinically significant or clinically significant. If abnormalities are observed, each will be recorded.

#### 7.2.9 Additional Data listings and tabulations

#### 7.2.9.1 Neurological Assessment

All neurological assessment results will be listed and any abnormality will be summarized.

### 7.2.9.2 Urine Pregnancy Test

All the results from urine pregnancy will be presented as a by-subject listing.

## 7.2.9.3 *Notification and Outcome Pregnancy*

All the results for Notification and Outcome Pregnancy will be presented as a by-subject listing.

7.2.9.4 HIV-1 Trofile® DNA/RNA Assay and Drug Resistance, Genotypic and Phenotypic data Data for HIV-1 trofile® DNA/RNA assay as well us Drug Resistance, Genotypic and Phenotypic data will be provided by external vendor Monogram Biosciences. All data will be presented as by-subject listings.

## 7.2.9.5 TruCount Assay (including CD4 Counts)

Data for TruCount assay will be provided by external vendor Covance. All data will be presented as by-subject listings.

# 8. APPENDIX 1: SCHEDULE OF ASSESSMENTS

# TABLE 1: SCHEDULE OF ASSESSMENTS – SCREENING AND TREATMENTPHASE

| Procedure/Assessments | Screening | Treatment Phase | | | | |
|---|---|---|---|---|---|---|
| Visit | Screening<br>(T23/24/25) | (EOT) | E1 <sup>b</sup> | Subsequent<br>TE Visits<br>(weekly ±3 days) | EOT | VF |
| | | Pre-treatment | Post-treatment | | | |
| Informed Consent <sup>[1]</sup> | Х | | | | | |
| Subject Demographics | Χ | | | | | |
| Medical & HIV History[2] | Χ | | | | | |
| Eligibility | Х | X | | | | |
| Physical Examination | X[3] | Χ | | X[3] | Χ | X[3] |
| Neurological Examination <sup>[4]</sup> | Χ | Χ | | | Χ | X |
| Vital Signs <sup>[5]</sup> | Χ | X | X | X | Χ | X |
| ECG | Χ | | | | X | |
| Complete Blood Count <sup>[6]</sup> | | Χ | | X <sup>[15]</sup> | Χ | Х |
| Biochemistry <sup>[7]</sup> | | Χ | | X <sup>[15]</sup> | Х | Х |
| Coagulation <sup>[8]</sup> | | Х | | X <sup>[15]</sup> | Х | Х |
| Urinalysis <sup>[9]</sup> | | Χ | | X <sup>[15]</sup> | Χ | Х |
| Urine pregnancy test <sup>[10]</sup> | | Х | | | | |
| Plasma HIV-1 RNA level[11] | Χ | Χ | | Х | Х | Х |
| TruCount T assay[11] | Χ | Х | | X | Х | Х |
| PRO 140 + OBT Regimen | Χ | ) | X . | X | Х | |
| Injection Site Reaction<br>Assessment -<br>Investigator <sup>[12]</sup> | Х | | х | х | Х | |
| HIV-1 Trofile <sup>®</sup> RNA +<br>PhenoSense Entry Assay <sup>[13]</sup><br>] | | | | | | х |
| HIV-1 Drug Resistance<br>Assay <sup>[14]</sup> | | | | | | х |
| Adverse Events | Χ | | Х | Х | Х | Х |
| Concomitant Medications | Х | Х | | Х | Х | Х |

- X (red bold with yellow highlight): Activities performed under PRO 140\_CD02 study protocol 
  <sup>a</sup> Schedule of assessment (Screening/Treatment Phase) can be modified by the Investigator based 
  on clinical judgment and in the best interest of the subject.
  - <sup>b</sup> Subject eligibility should be confirmed <u>prior</u> to study treatment administration at TE1.

#### Foot Notes:

- [1] Informed consent must be obtained prior to subject participation in any protocol-related activities that are not part of routine care.
- [2] Medical history, past surgeries, disease history, history of substance abuse, social history, blood transfusion history, and current therapies (medications and non-medications) will be brought forward from PRO140 CD02.
- [3] Symptom-directed physical examination. Complete physical examination at TE1, EOT2 and VF.
- [4] The screening tool for this assessment is based on the three question survey used by Simioni et al. (Simioni S, 2010). Additional modalities may be used for this assessment at the discretion of the Investigator.
- [5] Vital signs (i.e., blood pressure, heart rate, respiration rate and temperature) will be recorded posttreatment whenever IP administered at the clinic.
- [6] Hemoglobin, Hematocrit (HCT), Red Blood Cells (RBC), White Blood Cells (WBC) with total and differential count, Absolute Neutrophil Count (ANC) and platelets.
- [7] Serum Biochemistry

Hepatic function indicators: total and direct bilirubin, alkaline phosphatase, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total protein, Lactate dehydrogenase (LDH)

Renal function indicators: BUN, creatinine

Electrolytes: sodium, potassium, chloride, calcium and bicarbonate

Other: glucose (random), cholesterol (total)

- [8] Prothrombin time (PT) and International Normalized Ratio (INR)
- [9] Urine samples will be tested for color, appearance, specific gravity, pH, protein, glucose, occult blood, ketones, leukocyte esterase, nitrite, bilirubin, urobilinogen, and microscopic examination of urine sediment.
- [10] ONLY performed on women of childbearing potential. Subject will not be allowed to participate if the result is positive.
- [11] Plasma HIV-1 RNA and TruCount T Assay will be performed once every 4 weeks when subject comes to clinic. TruCount T Assay includes: CD3 %, CD4 %, CD8 %, Absolute Lymphocytes, CD3 cell count, CD4 cell count, and CD8 cell count
- [12] Injection Site Reaction will be assessed by the Investigator whenever IP administered at the clinic.
- [13] Monogram Biosciences Trofile® RNA and PhenoSense® Entry Assays [AMD3100 (CXCR4 inhibitor drug), Maraviroc and PRO 140 (CCR5 inhibitor drugs)]
- [14] Monogram Biosciences PhenoSense® GT Assay
- [15] Every 12 weeks during Treatment Extension.

## TABLE 8-2: SCHEDULE OF ASSESSMENTS - FOLLOW-UP (FU) PHASE

(a) Subjects who do NOT experience virologic failure

| Procedure/Assessments | Follow-Up Visit -1 | Follow-Up Visit -2 |
|---|---|---|
| | NVF-EFU1 | NVF-EFU2 |
| Window Period | 2 weeks<br>(±3 days) after EOT2<br>visit | 4 weeks<br>(±3 days) after EOT2 visit |
| Physical Examination | X <sup>[1]</sup> | χ[1] |
| Vital Signs | X | X |
| Plasma HIV-1 RNA level | X | X |
| TruCount T assay | X | X |
| Adverse Events | Х | X |
| Concomitant Medications | X | X |

<sup>[1]</sup> Symptom-directed physical examination

# (b) Subjects who experience virologic failure

| Procedure/Assessments | Follow-Up Visit -1 | Follow-Up Visit -2 | Follow-Up Visit -3 <sup>[1]</sup> |
|---|---|---|---|
| | VF-EFU1 | VF-EFU2 | VF-EFU3 |
| Window Period | 4 weeks<br>(±7 days) after VF<br>visit | 8 weeks<br>(±7 days) after VF | 12 weeks<br>(±7 days) after VF |
| Physical Examination | X[2] | χ[2] | Χ[2] |
| Vital Signs | X | X | X |
| Plasma HIV-1 RNA level | X | X | X |
| TruCount T assay | X | X | X |
| Adverse Events | X | X | X |
| Concomitant Medications | X | X | X |

<sup>[1]</sup> Subject will be followed up till the viral suppression is achieved or up to a maximum of 6 months after experiencing Virologic Failure (VF) if the treating physician does not feel that there is an antiretroviral regimen that will regain full viral suppression.

<sup>[2]</sup> Symptom-directed physical examination

#### 9. APPENDIX 2 - PLANNED TLG

# 9.1 Planned by-subject listings

DISPOSITION/WITHDRAWALS (LISTINGS 16.2.1.X)

ELIGIBILTY AND PROTOCOL DEVIATIONS (LISTINGS 16.2.2.X)

EXCLUDED SUBJECTS (LISTINGS 16.2.3.X)

DEMOGRAPHICS, POPULATION, AND BASELINE CHARACTERISTICS (LISTINGS 16.2.4.X)

TREATMENT ADMINISTRATION LISTINGS (LISTINGS 16.2.5.X)

EFFICACY RESPONSE DATA (LISTINGS 16.2.6.X)

ADVERSE EVENT DATA (LISTINGS 16.2.7.X)

SAFETY DATA (LISTINGS 16.2.8.1.X)

# 9.2 Planned Summary Tables

POPULATION DISPOSITION AND PROTOCOL DEVIATIONS
POPULATION DEMOGRAPHICS AND BASELINE CHARACTERISTICS
CONCOMITANT MEDICATION USAGE
EFFICACY SUMMARIES

**SAFETY SUMMARIES** 

ADVERSE EVENT SUMMARIES

SERIOUS ADVERSE EVENTS

LABORATORY

VITAL SIGNS AND PE

**OTHER SAFETY** 

#### 10 REFERENCES

- 1. ASA Ethical Guidelines for Statistical Practice (2016)
- 2. The Royal Statistical Society: Code of Conduct (2014)
- 3. ICH Guidance on the Structure and Content of Clinical Study Reports (ICH E3, 1996)
- 4. ICH Guidance on the Structure and Content of Clinical Study Reports (ICH E3(R1), 2013)
- 5. ICH Guidance on the Statistical Principles for Clinical Trials (ICH E9, 1998)
- 6. ICH Guidance on the Statistical Principles for Clinical Trials (ICH E9(R1), 2017)

| 1 | 1 | 1 | ZΕ | R | SI | $\mathbf{C}$ | N | $\mathbf{H}$ | IS | T | N | R | 1 | <b>Y</b> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

This is the first version of the document.